CLINICAL TRIAL: NCT04867122
Title: Problem-Solving Therapy for Cancer Caregivers: A Randomized Clinical Trial in Outpatient Palliative Care
Brief Title: Problem-Solving Therapy for Cancer Caregivers in Outpatient Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Pennsylvania (Other); National Cancer Institute (NCI) (NIH); University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202104120; R01CA258311 (NIH)
Record Dates: First submitted 2021-03-26; First posted 2021-04-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Depression, Anxiety; Palliative Care; Caregivers; Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: The randomized portion of the trial will enroll 540 family caregivers. An additional portion of the trial will enroll 30 key stakeholders to participate in individual interviews focused on potential barriers and facilitators to adoption of the problem-solving therapy (PST) intervention into clinical practice.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Attention Control (Placebo Comparator): Family caregivers in the attention control study arm will receive three sessions of attention-matched control in addition to the services and support provided as part of usual outpatient palliative care. Attention-matched control will consist of three "friendly visits" with a trained research staff person.
  Interventions: Other: Attention-matched Control
- Problem Solving Therapy Intervention (Experimental): Family caregivers in the intervention study arm will participate in three problem-solving therapy sessions with a trained interventionist in addition to receiving the services and support provided as part of usual outpatient palliative care.
  Interventions: Behavioral: Problem-Solving Therapy
- In-Depth Interviews for non-FCG Stakeholders (Other): Each year of the project, the investigators will recruit 6 key stakeholders to participate in individual interviews focused on potential barriers and facilitators to adoption of the PST intervention into clinical practice for a total of 30 unique stakeholders who will be interviewed over the duration of this 5-year study.
  Interventions: Other: In-depth interviews

INTERVENTIONS:
Behavioral: Problem-Solving Therapy — Over an approximately 3-week period, family caregivers randomized to the intervention study arm will learn and apply a problem-solving approach based on the ADAPT model, which encourages participants to follow five steps when solving caregiving problems: 1) focus on adopting a positive attitude to problem solving, 2) define the problem and set goals, 3) generate a list of alternative solutions to the problem, 4) predict consequences of the alternative solutions, and 5) try implementing the most promising solution from among the list of alternatives. The intervention will be delivered by a trained interventionist over the course of three structured sessions via telephone or videoconferencing technology, depending on the FCG's preference. Session content will be summarized in an intervention manual, which we will provide to all intervention participants. Sessions will last approximately 45-60 minutes.
  Arms: Problem Solving Therapy Intervention
Other: Attention-matched Control — Over an approximately 3-week period, family caregivers randomized to the attention control study arm will participate in informal conversations ("friendly visits") with a trained member of the research team.
  Arms: Attention Control
Other: In-depth interviews — The 30 key stakeholders interviews will discuss how the PST intervention fits into existing clinical practice and institutional values, what might incentivize adoption of the PST intervention, and how the intervention compares to alternative existing or proposed programs.
  Arms: In-Depth Interviews for non-FCG Stakeholders

SUMMARY:
This study is a randomized clinical trial of a problem-solving therapy intervention for family caregivers of individuals with cancer receiving outpatient palliative care.

DETAILED DESCRIPTION:
This study is a randomized clinical trial of a problem-solving therapy intervention for family caregivers of individuals with cancer receiving outpatient palliative care. Study participants will be randomized to receive either a three-session problem-solving therapy intervention in addition to usual care or three sessions of attention-matched control in addition to usual care.

ELIGIBILITY:
Inclusion Criteria for Family Caregivers (FCGs)

* Must be 18 years of age or older
* Must serve as the unpaid family caregiver of a patient with cancer receiving outpatient palliative care from one of the participating clinical sites. As is common in caregiving research, we will define "family caregiver" as anyone substantially involved in a patient's care on an unpaid basis; a legal or biological relationship will not be required
* Must consent to participate

Inclusion Criteria for Non-Family Caregiver Stakeholders

* Must be 18 years of age or older
* Must be employed by or affiliated with the healthcare system housing one of the participating clinical sites.
* Must consent to participate.

Exclusion Criteria for Family Caregivers (FCGs)

* Younger than 18 years of age
* Paid caregiver

Exclusion Criteria for Non-Family Caregiver Stakeholders

* Younger than 18 years of age
* Not employed by or affiliated with the healthcare system housing one of the participating clinical sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Change in anxiety as measured by the PROMIS Short Form v1.0 - Anxiety 8a | At the time of enrollment, Week 4, and 30-day follow-up
  Family caregivers indicate the frequency with which they experience eight different symptoms of anxiety (8 items); higher scores reflect higher anxiety severity.
Change in symptoms of depression as measured by the PROMIS Short Form v1.0 - Depression 8a | At the time of enrollment, Week 4, and 30-day follow-up
  Family caregivers indicate the frequency with which they experience eight different symptoms of depression (8 items); higher scores reflect higher depression severity

SECONDARY OUTCOMES:
Change in positive aspects of caregiving as measured by Positive Aspects of Caregiving Scale - Short Form (S-PAC; 7 items) | At the time of enrollment, Week 4, and 30-day follow-up
  * Family caregivers indicate good things that they experience as a caregiver with seven different statements. The caregivers answer with 1=I disagree with this statement a lot; 2=I disagree with this statement a little; 3=I neither agree nor disagree with this statement; 4=I agree with this statement a little; or 5=I agree with this statement a lot.
  * Higher scores indicate a more positive caregiving experience

CONTACTS AND LOCATIONS:
Overall Officials: Karla Washington, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - University of Missouri, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pennslyvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu